CLINICAL TRIAL: NCT00157118
Title: A Phase II/III Clinical Study for the Determination of the Efficacy and Safety of Protein C Concentrate in Subjects With Severe Congenital Protein C Deficiency
Brief Title: Efficacy and Safety Study of Protein C Concentrate in Subjects With Severe Congenital Protein C Deficiency
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 400101
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Protein C Deficiency
Keywords: Severe congenital protein C deficiency
MeSH Terms: conditions — Protein C Deficiency | interventions — Protein C

INTERVENTIONS:
Drug: Protein C Concentrate (Human) Vapor Heated

SUMMARY:
The purpose of this study is to show that Protein C Concentrate is a safe and effective treatment for subjects with congenital protein C deficiency. Depending on the type of treatment required, patients are assigned to one of 3 study parts: Part 1 is for the treatment of acute episodes, Part 2 is for short-term prophylaxis, and Part 3 is for long-term prophylaxis in infants aged less than 6 months only.

ELIGIBILITY:
Inclusion Criteria:

* Newborn subjects <= 6 months of age: diagnosis of severe congenital protein C deficiency, with documented functional protein C level < 20%. If a genetic diagnosis is not available prior to initiation of Protein C Concentrate treatment, a documented family history of protein C deficiency is required.
* Subjects > 6 months of age: confirmed diagnosis of severe congenital protein C deficiency, i.e., by
* a genetic analysis of severe congenital protein C deficiency (i.e., homozygous or double heterozygous) OR
* a documented family history of protein C deficiency AND a documented functional protein C level < 20% while the subject is in an asymptomatic state and not receiving oral anticoagulation therapy
* Signed and dated informed consent from either the subject or the subject's legally authorized representative prior to enrollment. Informed consent includes consent for conducting a genetic analysis (if the genetic defect is unknown).

Exclusion Criteria:

* Subjects with a history of allergic reactions to Protein C Concentrate. In the case of allergic reactions occurring at the Protein C Concentrate injection site; exclusion from the study is at the discretion of the investigator but should be reported as an AE regardless of the subject's inclusion in or exclusion from the study.
* Participation in any clinical study in which another investigational agent is used within 30 days prior to enrollment or its use is expected at any time for the duration of study participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-08-22 (Actual); Primary Completion 2005-03-17 (Actual); Study Completion 2005-03-17 (Actual)

PRIMARY OUTCOMES:
Whether episodes of purpura fulminans, Coumarin-induced skin necrosis and/or other thromboembolic event could be treated effectively, effectively with complications, or not treated effectively with Protein C Concentrate. | Part 1 of the study

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- United States (12):
  - Los Angeles, California
  - Denver, Colorado
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Fort Worth, Texas
  - Galveston, Texas
  - Houston, Texas

REFERENCES:
- [Result] Gelmont D., Hays T., Bomgaars L., Palascak J., Shapiro A., Geil J., Montgomery J., Fritsch S., Maritsch F., Pavlova B., Ehrlich H.J. A Phase II/III Clinical Study for the Determination of the Efficacy and Safety of Protein C Concentrate in Subjects with Severe Congenital Protein C Deficiency -Interim Study Analysis. Accepted for poster presentation at the 20th International Society on Thrombosis and Haemostasis Congress. Sydney, Australia, August 6-12 2005. (ISTH 2005)